CLINICAL TRIAL: NCT05730764
Title: A Prediction Model and Assisted Decision-making System of Fertilization Disorders: a Single-center Randomized Controlled Trial
Brief Title: A Prediction Model and Assisted Decision-making System of Fertilization Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00006761-M2022487
Record Dates: First submitted 2023-01-16; First posted 2023-02-16 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2022-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Support systems assist doctors in decision-making (Experimental): Doctors judge the risk of fertilization disorders and make clinical decisions with the support of a decision-making system.
  Interventions: Diagnostic Test: Accurate prediction of fertilization disorders and clinical decision support systems assist doctors in decision-making
- Clinicians follow a routine protocol (Other): Doctors judge the risk of fertilization disorders and make clinical decisions based on clinical experience
  Interventions: Diagnostic Test: Clinicians follow a routine protocol

INTERVENTIONS:
Diagnostic Test: Accurate prediction of fertilization disorders and clinical decision support systems assist doctors in decision-making — With the assistance of accurate prediction of fertilization disorders and clinical decision support systems, clinicians predict and judge the probability and key factors of fertilization disorders of patients, and formulate and implement personalized diagnosis and treatment plans based on the prediction results
  Arms: Support systems assist doctors in decision-making
Diagnostic Test: Clinicians follow a routine protocol — Treatment is performed by the clinician according to the usual protocol.
  Arms: Clinicians follow a routine protocol

SUMMARY:
The goal of this clinical trial is to test the accuracy of the forecasting system we develop. The main question it aims to answer is:

* Whether the clinical prediction system predicts the incidence of fertilization disorders accurately.
* The fertilization disorder prediction system predicts whether and how much the outcome differs from the doctor.

Participants will receive treatment assisted by a predictive system or receive general treatment.

Researchers will compare incidence of fertilization disorders to see if the fertilization disorder prediction system makes correct predictions.

DETAILED DESCRIPTION:
Through the design method of single-center randomized controlled trial, 260 infertility patients were recruited, and they were divided into two groups of 130 cases in each group according to the method of block randomization, one of which was the intervention group, with the help of accurate prediction of fertilization disorders and clinical decision support systems, clinicians predicted and judged the probability and key factors of fertilization disorders of patients, and formulated and implemented personalized diagnosis and treatment plans based on the prediction results; The other group is the control group, which is treated by clinicians according to the conventional diagnosis and treatment plan, and the system performs parallel simulation operation to predict the outcome of fertilization disorders in patients without affecting any diagnosis and treatment decisions of clinicians. Through the comparison of the two groups, the predictive ability of the system for fertilization disorders was evaluated, and the effectiveness and safety of the personalized diagnosis and treatment plan formulated with the assistance of the system were observed, the primary observation outcomes were the incidence of fertilization disorders, and the secondary observation outcomes were embryo transfer rate, biochemical pregnancy rate, clinical pregnancy rate, etc.

ELIGIBILITY:
Inclusion Criteria:

1. infertile couples
2. have indications for acceptance of IVF or ICSI
3. Both parties sign an informed consent form and can complete the follow-up visit

Exclusion Criteria:

1. At least one of the spouses has contraindics to IVF or ICSI
2. Major diseases
3. Fresh cycle, PGT, IVM

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of fertilization disorders | through study completion, an average of 3 months
  Occurrence of fertilization disorders in participants

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China